CLINICAL TRIAL: NCT00829686
Title: Prospective Randomized Controlled Trial of Antibiotic Treatment for Uncomplicated Skin Abscess in Patients at Risk for Community Acquired Methicillin-Resistant Staphylococcus Aureus Infection
Brief Title: Trial of Antibiotic Treatment for Skin Abscess in Patients at Risk for Methicillin-Resistant Staphylococcus Aureus (MRSA) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gillian Schmitz, PI, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20080055H-Pilot
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Abscess
Keywords: abscess; cellulitis; antibiotics; MRSA
MeSH Terms: conditions — Abscess; Cellulitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention): No antibiotic
- Septra DS (Active Comparator): Septra DS (800/160) two pills PO BID x 7 days
  Interventions: Drug: Septra

INTERVENTIONS:
Drug: Septra — (800/125) PO BID X 7 days
  Arms: Septra DS

SUMMARY:
Patients will be enrolled in a multi-center study to prospectively evaluate outcome after treatment for an uncomplicated skin abscess. All patients will receive incision and drainage and wound cultures. Patients will then be randomized to 1)no antibiotic or 2) bacterium double strength (DS) (800/160) two tablets per oral (PO) twice a day x 7 days. This is the dose recommended for treating skin and soft tissue infections. (Ellis et al. Current Opinion in Infectious Diseases. 18(6):496-501, December 2005) Patients will then return to the emergency room (ER) on days 3 and 7 for wound repacking and evaluation. The primary outcome is clinical cure of abscess at 7 days after incision and drainage and recurrence rates within 30 days of treatment. Patients who are not improving at the following visit will then be treated with additional antibiotics or admission if needed. Data will be analyzed both by initial randomization and intention to treat. This serves as the pilot for the full placebo controlled randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* all patients age 18-55 who present to the emergency department with a skin abscess that requires incision and drainage.

Exclusion Criteria:

* patients with diabetes, HIV, cancer or other immunocompromised patients
* patients who received antibiotics within one week of presentation or were hospitalized in previous month will be excluded to minimize potential confounding variables
* pregnant and breastfeeding patients will also be excluded due to possible safety concerns with antibiotic treatment
* basic Military Trainees will also be excluded from participation
* patients with abscesses on head, face, perirectal, or periananal regions, abscesses with known tracks or fistulas to deeper structures, or abscesses requiring surgical drainage in an operating room are excluded
* patients with sulfa allergy will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilford Hall Medical Center, Lackland Air Force Base, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited who presented to the ER with an uncomplicated skin abscess who met inclusion criteria and did not meet exclusion criteria. Informed consent was obtained.
Period: Overall Study
Arm/Group | No Intervention | Septra DS
Started | 13 | 18
Completed | 13 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Septra DS | Total
Number analyzed (Participants) | 13 | 18 | 31
Age, Categorical [Count of Participants; unit: Participants] — Age (Years)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 13 | 18 | 31
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (2) | 34.5 (2) | 34.3 (2)
Age, Customized [Count of Participants; unit: Participants]
  Age 18-25 years | 6 | 7 | 13
  Age 26-40 years | 2 | 3 | 5
  Age 41-65 years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement at 7 Days After Incision and Drainage
Description: improving wound without evidence of fever, worsening cellulitis or induration
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | No Intervention | Septra DS
Number analyzed (Participants) | 13 | 18
participants | 10 | 14

2. Secondary Outcome: Recurrence Rates
Description: recurrence of abscess in previous or new location within 30 days
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | No Intervention | Septra DS
Number analyzed (Participants) | 13 | 18
participants | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No